CLINICAL TRIAL: NCT01931813
Title: Pharmacoepidemiological Methodology to Evaluate the Vaccination Risk in Young Infants
Brief Title: METHORIVAC - Vaccinal Pharmacoepidemiologic
Acronym: METHORIVAC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Quantin PHRC IR 2009
Record Dates: First submitted 2013-08-27; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Infants Likely to Present Febrile Convulsions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants likely to present febrile convulsions

SUMMARY:
This project is the pilot step necessary to develop a system of vaccination pharmacoepidemiology that associates a sophisticated analytical approach, appropriate for this challenge and case series analysis, with the use of linked medicoadministrative data for hospitalisations the reimbursement of healthcare costs. This linkage of medicoadministrative data is new in France. The example of the risk of hospitalisation for febrile convulsions in infants less than two years old following vaccination against diphtheria, tetanus and pertussis is given as the reference association. This choice is justified by the numerous publications over many years on the existence of this association (Miller et al BMJ 1981, Farrington et al Lancet 1995). In addition, as case series analyses have been carried out to assess this risk, the results can be compared directly (Lancet 1995). The study to determine whether the analysis tools are suitable for the data will be tackled at the following levels:

* Validity of the selection of cases from administrative records alone using coding based on the international classification of diseases ICD10
* Validity of the risk assessment. This methodology feasibility project must make it possible to identify the different potential problems. This is a prerequisite necessary for the systematic implementation.

ELIGIBILITY:
Inclusion Criteria:

- For reimbursement data: All of the data concerning delivery (purchase of the vaccine at a pharmacy, prescription) and vaccination (consultation following the date of purchase) for infants younger than 2 years old, in the years 2007 and 2008.

- For PMSI data: All of the hospitalisations in 2007 and 2008 for febrile convulsions in infants less than 3 years old in hospitals of the following departments: Côte d'Or, Doubs and Bas-Rhin

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children of less than 3 years hospitalized for febrile convulsions
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
DATA EXTRACTION | At the selection of patients
  Dates of delivery (purchase of the vaccine at the pharmacy), prescription, and date of vaccination (consultation) and when necessary, the age, doses, dates of adverse events, identification of the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France